CLINICAL TRIAL: NCT02953912
Title: Assessment of Postoperative Pain After Using Reciproc Versus One Shape NiTi Systems in Patients With Symptomatic Irreversible Pulpitis.
Brief Title: Assessment of Postoperative Pain Using Reciproc Versus One Shape Files in Patients With Irreversible Pulpitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Kamal, principal investigator., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: reciproc_one shape
Record Dates: First submitted 2016-10-31; First posted 2016-11-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-10

CONDITIONS: Pulpitis - Irreversible
Keywords: Rotation; Reciprocation; single file; postoperative pain; Reciproc; One Shape; Symptomatic irreversible pulpitis
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reciproc single-file. (Experimental): The Reciproc is a single-file nickel-titanium systems used in reciprocating motion, made of a special nickel-titanium (NiTi) alloy called M-Wire created by innovated thermal treatment process which increases flexibility and improved resistance to cyclic fatigue .
  Interventions: Procedure: Reciproc single-file
- One Shape single-file . (Active Comparator): One Shape is single file made of austenite 55- NiTi alloy characterized by different cross sectional designs ,it is used in continuous clockwise rotation for a quick and safe root canal preparation due to its flexibility and minimal fatigue. with electropolished safety tip instrument for enhanced cutting efficiency and it is delivered in a sterile blister for single use.
  Interventions: Procedure: One Shape single-file

INTERVENTIONS:
Procedure: Reciproc single-file — The Reciproc is a single-file nickel-titanium systems , made of a special nickel-titanium (NiTi) alloy called M-Wire created by innovated thermal treatment process which increases flexibility and improved resistance to cyclic fatigue
  Arms: Reciproc single-file.
Procedure: One Shape single-file — One Shape is one of the few single file made of austenite 55- NiTi alloy characterized by different cross sectional designs ,it is used in continuous clockwise rotation for a quick and safe root canal preparation due to its flexibility and minimal fatigue.In addition to , the electropolished safety tip instrument for enhanced cutting efficiency and it is delivered in a sterile blister for single use.
  Arms: One Shape single-file .

SUMMARY:
To show whether One Shape rotary system differs from Reciproc reciprocating system in postoperative pain in patients with symptomatic irreversible pulpitis.

DETAILED DESCRIPTION:
Patients in the clinic of endodontics at the faculty of oral and dental medicine, Cairo University, Urban area, Cairo governorate, Egypt.

The dental Unit is Adec 200 U.S.A. The x-ray Machine is ViVi, S.r.I, Italy The x-ray films are Kodac, speed D, size 2. The operator is master degree student in the department of Endodontics. No dental assistant Time: 2016-2017 Diagnosis The diagnostic data will be collected in a case report form by the investigator and confirmed for eligibility with the assistant supervisor and will be enrolled in the study in the same day.

Diagnosis is done by the following:

Recording the chief complaint and history of pain Clinical examination will be evaluated for (sensitivity) of pulp tissues using cold testing (by using Green Endo ice), electric tester.

The patient should experience prolonged response to cold testing and positive response to electric pulp testing Radiographic examination: There should be no periapical radiolucency except for widening periodontal ligaments.

Intervention Full medical and dental history using a schematic dental chart will be obtained from all patients treated during this study. Each tooth will be evaluated for vitality (sensitivity) of pulp tissues using electric pulp tester.

The patients will be randomly divided into 2 group:

Experimental group Reciproc single-file reciprocating instrumentation system. Control group One Shape single-file rotary instrumentation system. Sequence of Procedural steps Preoperative pain will be assessed by NRS before administration of anesthesia. Local anesthesia will be achieved using 2% lidocaine (1:100,000 adrenaline). An access cavity will be performed using round bur and Endo-Z bur1.

. The tooth will be properly isolated with rubber dam. Working length will be determined using an electronic apex locator2, and working length will be confirmed by radiograph using K-file3. Then the working length will be established at 0.5 mm up to the radiographic apex.

Canals will be explored with hand K-file ISO sizes 10, 15, 20. Mechanical preparation for both groups will be as follows

Experimental group Canals will be instrumented using Reciproc4 reciprocating system set on an electric motor5, with adjusted torque and speed according to the manufacturer's instruction.

There is no need for coronal preflaring with a Gates Glidden drill or an orifice opener since the design of the Reciproc instrument allows any obstructions in the coronal third to be removed, as claimed by the - Reciproc file selection: R40 (40/0.06) manufacturer.

Control group Coronal preflaring will be performed using Gates Glidden drill. Canals will be instrumented using One Shape1 single-file (25/0.06) set on an electric motor2 with adjusted torque and speed according to the manufacturer's instructions.

For wide canals, One Shape Apical (30/0.06, 37/0.06) will be used. The rotary files will be introduced inside the canal using EDTA gel3.. Canals will be irrigated with 2.5% sodium hypochlorite solution between every subsequent instrument. It is prepared by adding 11 ml of sterile distilled water using a 27 gauge needle fit to 5ml disposable plastic syringe placed in the canal space without binding

Canals will be dried with sterile paper points and obturated using lateral condensation technique. A spreader will be used to allow space for auxiliary cones, with resin-based root canal sealer.

The tooth will be sealed by temporary restoration, and postoperative pain will be assessed immediately after the end of treatment.

The patient will be phone called for follow up after 6, 12, 24, 48 and 72 hours.

The patient will be instructed to return to complete the treatment procedures until placing a full-coverage restoration.

The patient will be instructed to take one tablet 600 mg Ibuprofen if he/she experiences severe pain.

Outcomes Primary Outcome :Intensity of postoperative pain will be measured using a numerical rating scale (NRS) immediately after the end of treatment, 6, 12, 24, 48, and 72 hours after the end of endodontic treatment.

The numerical rating scale (0-10 scale) consists of a line anchored by two extremes "0: no pain" and "10: severe pain"; patients will be asked to choose the mark that represents their level of pain from 0 to 10. Pain level will be assigned to one of 4 categorical scores:

0, None; 1, Mild (1-3); 2, Moderate (4-6); 3, Severe (7-10)

0: None

1. Mild (1-3)
2. Moderate (4-6)
3. Severe (7-10)

Secondary outcome Number of analgesic taken by the patient to decrease postoperative pain up to 3 days after the end of endodontic treatment will be recorded by the patient with time intervals.

Participant Timeline:

After the patient is found eligible, he/she will be randomly assigned to either the control (One Shape) or experimental group (Reciproc) and will be treated in a single visit. At the end of treatment, patients will be asked to record postoperative pain by NRS immediately, then after 6,12,24,48 and 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* i. Age 25-45years old. ii. Males or Females. iii. Mandibular premolar teeth with:

  * Single canal
  * Preoperative sharp pain.
  * Vital response of pulp tissue.
  * Normal periapical radiographic appearance or slight widening in lamina dura.

Exclusion Criteria:i. Patients who have already consumed preoperative medication, such as analgesic, non-steroidal or steroidal anti-inflammatory drugs, within 12 hours before treatment.

ii. Patients who have more than one tooth in the same quadrant and/or opposite quadrant that require an endodontic treatment.

iii. Pregnant females. iv. Patients having significant systemic disorder. v. If antibiotics have been administrated during the past two weeks preoperatively.

vi. Patients having bruxism or clenching. vii. Teeth that have:

* Non-vital pulp tissues.
* Association with swelling or fistulous tract.
* A pocket depth greater than 5 mm.
* Previous endodontic treatment.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-10 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain after endodontic treatment | immediately after the end of treatment up to 72 hours
  Intensity of postoperative pain will be measured using a numerical rating scale (NRS)

SECONDARY OUTCOMES:
Number of analgesic tablets taken by the patient after endodontic treatment | Within 3 days after endodontic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa I Gawdat, Lecturer, Study Director — Department of endodontics - Faculty of Oral and Dental medicine - CU; Angie G Ghoneim, Professor, Study Chair — Department of endodontics - Faculty of Oral and Dental medicine - CU; Asmaa M kamel, Student, Principal Investigator — Department of endodontics - Faculty of Oral and Dental medicine - CU

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sathorn C, Parashos P, Messer H. The prevalence of postoperative pain and flare-up in single- and multiple-visit endodontic treatment: a systematic review. Int Endod J. 2008 Feb;41(2):91-9. doi: 10.1111/j.1365-2591.2007.01316.x. Epub 2007 Oct 23. PMID 17956561
- [Background] Gondim E Jr, Setzer FC, Dos Carmo CB, Kim S. Postoperative pain after the application of two different irrigation devices in a prospective randomized clinical trial. J Endod. 2010 Aug;36(8):1295-301. doi: 10.1016/j.joen.2010.04.012. Epub 2010 Jun 19. PMID 20647083
- [Background] Neelakantan P, Sharma S. Pain after single-visit root canal treatment with two single-file systems based on different kinematics--a prospective randomized multicenter clinical study. Clin Oral Investig. 2015 Dec;19(9):2211-7. doi: 10.1007/s00784-015-1448-x. Epub 2015 Mar 15. PMID 25773449
- [Background] Shuping GB, Orstavik D, Sigurdsson A, Trope M. Reduction of intracanal bacteria using nickel-titanium rotary instrumentation and various medications. J Endod. 2000 Dec;26(12):751-5. doi: 10.1097/00004770-200012000-00022. PMID 11471648
- [Background] Nekoofar MH, Sheykhrezae MS, Meraji N, Jamee A, Shirvani A, Jamee J, Dummer PM. Comparison of the effect of root canal preparation by using WaveOne and ProTaper on postoperative pain: a randomized clinical trial. J Endod. 2015 May;41(5):575-8. doi: 10.1016/j.joen.2014.12.026. Epub 2015 Feb 24. PMID 25720984
- [Background] Siqueira JF Jr, Rocas IN, Favieri A, Machado AG, Gahyva SM, Oliveira JC, Abad EC. Incidence of postoperative pain after intracanal procedures based on an antimicrobial strategy. J Endod. 2002 Jun;28(6):457-60. doi: 10.1097/00004770-200206000-00010. PMID 12067129
- [Background] Tinaz AC, Alacam T, Uzun O, Maden M, Kayaoglu G. The effect of disruption of apical constriction on periapical extrusion. J Endod. 2005 Jul;31(7):533-5. doi: 10.1097/01.don.0000152294.35507.35. PMID 15980716
- [Background] Seltzer S, Naidorf IJ. Flare-ups in endodontics: I. Etiological factors. J Endod. 1985 Nov;11(11):472-8. doi: 10.1016/S0099-2399(85)80220-X. No abstract available. PMID 3868692
- [Background] Harrington GW, Natkin E. Midtreatment flare-ups. Dent Clin North Am. 1992 Apr;36(2):409-23. PMID 1572507
- [Background] Munoz E, Forner L, Llena C. Influence of operator's experience on root canal shaping ability with a rotary nickel-titanium single-file reciprocating motion system. J Endod. 2014 Apr;40(4):547-50. doi: 10.1016/j.joen.2013.08.027. Epub 2013 Oct 13. PMID 24666909
- [Background] Peters OA, Schonenberger K, Laib A. Effects of four Ni-Ti preparation techniques on root canal geometry assessed by micro computed tomography. Int Endod J. 2001 Apr;34(3):221-30. doi: 10.1046/j.1365-2591.2001.00373.x. PMID 12193268
- [Background] Ruddle CJ, Machtou P, West JD. The shaping movement: fifth-generation technology. Dent Today. 2013 Apr;32(4):94, 96-9. No abstract available. PMID 23659098
- [Background] Ferraz CC, Gomes NV, Gomes BP, Zaia AA, Teixeira FB, Souza-Filho FJ. Apical extrusion of debris and irrigants using two hand and three engine-driven instrumentation techniques. Int Endod J. 2001 Jul;34(5):354-8. doi: 10.1046/j.1365-2591.2001.00394.x. PMID 11482718
- [Background] Azar NG, Ebrahimi G. Apically-extruded debris using the ProTaper system. Aust Endod J. 2005 Apr;31(1):21-3. doi: 10.1111/j.1747-4477.2005.tb00202.x. PMID 15881729
- [Background] Burklein S, Benten S, Schafer E. Shaping ability of different single-file systems in severely curved root canals of extracted teeth. Int Endod J. 2013 Jun;46(6):590-7. doi: 10.1111/iej.12037. Epub 2012 Dec 13. PMID 23240965
- [Background] Park H. A comparison of Greater Taper files, ProFiles, and stainless steel files to shape curved root canals. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2001 Jun;91(6):715-8. doi: 10.1067/moe.2001.114159. PMID 11402288
- [Background] Burklein S, Schafer E. Apically extruded debris with reciprocating single-file and full-sequence rotary instrumentation systems. J Endod. 2012 Jun;38(6):850-2. doi: 10.1016/j.joen.2012.02.017. Epub 2012 Apr 6. PMID 22595125
- [Background] Yared G. Canal preparation using only one Ni-Ti rotary instrument: preliminary observations. Int Endod J. 2008 Apr;41(4):339-44. doi: 10.1111/j.1365-2591.2007.01351.x. Epub 2007 Dec 12. PMID 18081803
- [Background] Nabeshima CK, Caballero-Flores H, Cai S, Aranguren J, Borges Britto ML, Machado ME. Bacterial removal promoted by 2 single-file systems: Wave One and One Shape. J Endod. 2014 Dec;40(12):1995-8. doi: 10.1016/j.joen.2014.07.024. Epub 2014 Aug 19. PMID 25149120
- [Background] Capar ID, Arslan H. A review of instrumentation kinematics of engine-driven nickel-titanium instruments. Int Endod J. 2016 Feb;49(2):119-35. doi: 10.1111/iej.12432. Epub 2015 Feb 18. PMID 25630977
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Labbaf H, Shakeri L, Orduie R, Bastami F. Apical Extrusion of Debris after Canal Preparation with Hand-Files Used Manually or Installed on Reciprocating Air-Driven Handpiece in Straight and Curved Canals. Iran Endod J. 2015 Summer;10(3):165-8. doi: 10.7508/iej.2015.03.004. Epub 2015 Jul 1. PMID 26213538